CLINICAL TRIAL: NCT05107778
Title: A Phase II Multi-center, Randomized, Single-blind, Placebo-controlled to Evaluate Safety and Efficacy of ASC42 Tablets in Combination With Entecavir and Pegylated Interferon α-2a in Subjects With Chronic Hepatitis B Virus
Brief Title: Study to Evaluate Safety and Efficacy of ASC42 Combined With ETV and PEG-IFN α-2a in Subjects With HBV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASC42-201
Record Dates: First submitted 2021-10-26; First posted 2021-11-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; ASC42
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Queue ASC42 10mg (Experimental): ASC42 10mg, ih PEG-IFN α-2a and ETV for 12 weeks.
  Interventions: Drug: ASC42 10mg; Drug: ih PEG-IFN α-2a; Drug: Entecavir
- Queue ASC42 15mg (Experimental): ASC42 15mg , ih PEG-IFN α-2a and ETV for 12 weeks.
  Interventions: Drug: ASC42 15mg; Drug: ih PEG-IFN α-2a; Drug: Entecavir
- Queue Placebo (Placebo Comparator): Placebo, ih PEG-IFN α-2a and ETV for 12 weeks.
  Interventions: Drug: ih PEG-IFN α-2a; Drug: Entecavir; Drug: Placebo

INTERVENTIONS:
Drug: ASC42 10mg — ASC42 10mg orally once daily;
  Arms: Queue ASC42 10mg
Drug: ASC42 15mg — ASC42 15mg orally once daily.
  Arms: Queue ASC42 15mg
Drug: ih PEG-IFN α-2a — ih PEG-IFN α-2a 180μg subcutaneous injection once a week.
Drug: Entecavir — Entecavir 0.5 mg orally once daily.
Drug: Placebo — Placebo orally once daily.
  Arms: Queue Placebo

SUMMARY:
This is a phase2, randomized, single-blind, placebo controlled and multi-center study in adults with chronic hepatitis B virus. The study is aimed at evaluating efficacy and safety of ASC42 in combination with entecavir and pegylated interferon α-2a in subjects with chronic hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old (including 18 and 65 years old);
* Chronic HBV infection confirmed by serological, etiological and clinical diagnosis (HBsAg positive for more than 6 months);
* HBV-DNA negative after nucleoside (acid) treatment;
* Laboratory test values meet the following requirements :

  * Liver function : AST, ALT ≤ 3×ULN; serum total bilirubin≤2×ULN; direct bilirubin≤1.5×ULN; serum albumin≥35 g/L (blood collection is not within 2 weeks before transfusion of albumin);
  * Hematology: white blood cell count>3.0×109/L, ANC>1.5×109/L; platelet>1×ULN; hemoglobin 120g/L. (No blood transfusion (including transfusion of red blood cells and platelets) and EPO, TPO, leukocyte-stimulating factor were required within 2 weeks before blood collection) ;
  * Renal function: serum creatinine≤1×ULN;
  * Thyroid function: TSH and T4 in normal range or thyroid function can be completely controlled ;
  * Determination of serum immunoglobulin : IgM≤ULN;
  * Coagulation function: International normalized ratio: INR≤1×ULN;

Exclusion Criteria:

* Chronic HBV with unexplained portal hypertension;
* Subjects with liver cancer or serum AFP >1×ULN;
* Previously received FXR therapy;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Serum HBsAg change compared with baseline | Week 12 of intervention\Week 24 of follow-up
Serum HBV pgRNA change compared with baseline | Week 12 of intervention\Week 24 of follow-up

SECONDARY OUTCOMES:
Serum HBsAg change compared with baseline | Week 2, 4 ,8 of intervention\Week 4,12 of follow-up
Serum HBV pgRNA change compared with baseline | Week 2, 4 ,8 of intervention\Week 4,12 of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China